CLINICAL TRIAL: NCT05559112
Title: Effects of Vitamin D-Enriched Mushrooms on Vitamin D Status and Immune Function in Adults
Brief Title: Effects of Vitamin D-Enriched Mushrooms on Vitamin D Status and Immune Function and Inflammatory Status in Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Principal Investigator, Purdue University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: IRB-2022-750
Record Dates: First submitted 2022-09-26; First posted 2022-09-29 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Vitamin D Deficiency
Keywords: Mushroom; Immune function; Vitamin D2; randomized controlled trial
MeSH Terms: conditions — Vitamin D Deficiency

STUDY DESIGN:
Intervention Model Description: For this investigator-blinded, randomized, parallel design study, 50 participants (40 to finish; n=20/group) will complete a 12-week study period in which participants consume 84 g of vitamin-D enriched mushrooms containing 800 IU/serving or study powder (control) in the context of their usual diet. To assess the effects of including vitamin D-enriched mushrooms as part of participants' usual eating pattern on serum vitamin D status and indices of immune function and inflammatory status, we will measure circulating concentrations of 25-hydroxy-vitamin D2, pro- and anti-inflammatory cytokines, and immunoglobulins, among other immunity/inflammation outcomes. Health questionnaires related to perceived anxiety/depression and wellbeing are included to complement the currently funded longitudinal feeding study which includes these exploratory outcomes.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mushrooms (Experimental): Participants will consume their usual, unrestricted, self-selected diet plus 84 g of vitamin D-enriched mushrooms twice daily for 12 weeks.
  Interventions: Other: Vitamin D-enriched mushrooms
- No Mushrooms (Placebo Comparator): This is a behavioral control where no change in Vitamin D status is expected to occur. Participants will consume their usual, unrestricted, self-selected diet plus 1 tsp of dried study powder twice daily for 12 weeks.
  Interventions: Other: Study Powder

INTERVENTIONS:
Other: Vitamin D-enriched mushrooms — Participants will consume their usual, unrestricted, self-selected diet plus 84 g of vitamin D-enriched mushrooms twice daily (for a total of 168g per day) for 12 weeks.
  Arms: Mushrooms
Other: Study Powder — Participants will consume their usual, unrestricted, self-selected diet plus 1 tsp of dried study powder twice daily (2 tsp total per day) for 12 weeks. Study powder is a commercially available carbohydrate.
  Arms: No Mushrooms

SUMMARY:
We propose to assess the effects of including vitamin D-enriched mushrooms as part of participants' usual eating pattern primarily on 25(OH) vitamin D2 status and secondarily on immune function and inflammatory status.

DETAILED DESCRIPTION:
We hypothesize that consuming vitamin D-enriched mushrooms daily for 12 weeks will prevent decreases in serum 25-hydroxy-vitamin D2 concentrations. Secondarily, we hypothesize consuming vitamin D-enriched mushrooms daily for 12 weeks will improve clinical indicators of inflammatory status and alter/enhance immune status and immune cell function. This short-term randomized, controlled trial will provide important data to inform the plausibility, focus, and design of longer-term intervention trials, consistent with The Mushroom Council's research agenda regarding health-promoting effects of vitamin D-enriched mushrooms.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 25.0-34.9 kg/m^2
* Total cholesterol <240 mg/dL
* low density lipoprotein cholesterol < 160 mg/dL
* triglycerides <300 mg/dL
* fasting glucose < 110 mg/dL
* systolic/diastolic blood pressure < 140/90 mmHg
* body weight stable for 3 months prior (+- 3 kg)
* stable physical activity regiment 3 months prior
* medication use stable for 6 months prior
* non-smoking
* non-diabetic
* not acutely ill
* females not pregnant or lactating
* willing to refrain from taking vitamin D supplements or any supplements containing vitamin D
* No history of bariatric surgery
* Not extremely or severely depressed (Beck's Depression Inventory Score <= 30)
* Agree not to donate blood for at least one month prior to, during, and for one month after the study
* Agree not to travel to sunny locations during the study period
* Agree to forgo any tanning bed or other tanning procedures during the study
* Willing and able to consume mushrooms and travel to testing facilities

Exclusion Criteria:

* Age <30 or >70
* BMI <25 or >35kg/m2
* Total cholesterol >240 mg/dL, low-density lipoprotein cholesterol >160 mg/dL, triglycerides >300mg/dL, fasting glucose >110 mg/dL
* Systolic/diastolic blood pressure >140/90 mm Hg
* Body weight changes in previous 3 months (±3 kg)
* Changes in physical activity regimen in the previous 3 months
* Medication changes in the previous 6 months
* Extremely or severely depressed (Beck's Depression Inventory Score >30)
* Unwilling to refrain from taking vitamin D supplements or any supplements containing vitamin D
* Regiment of megadosing vitamin D
* Unwilling to not to travel to sunny locations during the study period
* Unwilling to forgo any tanning bed or other tanning procedures during the study
* History of bariatric surgery
* Consuming a restricted diet (such as keto, gluten free, high protein, low carb, etc.)
* Smoking
* Diabetic
* Acute illness
* Females pregnant or lactating
* Unwilling to not to donate blood for at least one month prior to, during, and for one month after the study
* Allergic to mushrooms or bread

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Change in serum 25-hydroxy-vitamin D2 concentration | 12 weeks
  25(OH) Vitamin D2/D3 by LC/MS

SECONDARY OUTCOMES:
Change in immunity/inflammation markers | 12 weeks
  Immunoglobulin G, Immunoglobulin A, Immunoglobulin M (mg/dL)
Change in immunity/inflammation markers | 12 weeks
  High Sensitivity C Reactive Protein (hs-CRP)
Change in immunity/inflammation markers | 12 weeks
  Cytokine 13 Panel (pg/mL)
Change in bone remodeling | 12 weeks
  Osteocalcin
Change in serum calcium concentrations | 12 weeks
  Parathyroid hormone (PTH)
Change in perceived depression from baseline to mid to post-intervention | 12 weeks
  Beck's Depression Inventory questionnaire
Change in perceived anxiety from baseline to mid to post-intervention | 12 weeks
  Patient Health Questionnaire-9
Change in cognitive function from baseline to mid to post-intervention | 12 weeks
  Repeatable Battery for the Assessment of Neuropsychological Status
Change in perceived daily mood from baseline to mid to post-intervention | 12 weeks
  Profile of Mood States
Change in perceived quality of life from baseline to mid to post-intervention | 12 weeks
  Medical Outcomes Study 36-Item Short Form Health Survey Version 2
Risk factors for cardiovascular disease | 12 weeks
  Complete metabolic panel
Risk factors for cardiovascular disease | 12 weeks
  Blood pressure
Risk factors for cardiovascular disease | 12 weeks
  Lipoprotein Particle Plus (LPP+) Panel
Risk factors for cardiovascular disease | 12 weeks
  Complete blood count (CBC)
Risk factors for type 2 diabetes | 12 weeks
  Complete metabolic panel
Body weight | 12 weeks
  Measures of weight (kg)

CONTACTS AND LOCATIONS:
Overall Officials: Wayne Campbell, Principal Investigator — Purdue University
Locations (1):
- Purdue University, Department of Nutrition Science, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: Undecided